CLINICAL TRIAL: NCT04287699
Title: The Effect of Labor Dance on Traumatic Birth Perception and Comfort
Acronym: labordance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bihter Akın, Asisstant Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Labor Dance
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Labor Pain; Fear of Childbirth
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The study was planned as randomized controlled. Pregnant women and their accompanying persons assigned to the study group will be informed about working in the tram room where the pregnant woman is before the active phase begins 'Using the Birth Dance Practice Guide (Annex 3) and cervical dilatation 4 cm. they will be asked to practice in accordance with this guide. Details of the application (such as dance time, rest time) will be recorded in the 'Birth Dance Control Guide' (Annex 4) by the researcher. Pregnant women will be followed by the doctor and midwife responsible for the pregnancy during the tram, and the researcher will not be involved in tram follow-up of the pregnant woman (cervical dilation, pediatric heart sound, contraction follow-up, vital signs of the pregnant woman).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- labor dance group (Experimental): The pregnant women and their spouses/partners who wanted to perform the practice were asked to inform the researcher when the labor started. The researcher stayed with the pregnant women and their spouses during the practice and labor process. The pregnant women started to dance with their spouses during the active phase of the labor process accompanied by meditation music in a dim, silent environment.The pregnant women started to dance with their spouses during the active phase of the labor process accompanied by meditation music in a dim, silent environment. The spouse or partner massaged the pregnant woman's sacral area while dancing.
  Interventions: Other: labor dance
- Control group (No Intervention): Only routine practices were performed with the control group, and data were recorded as in the experimental groups.

INTERVENTIONS:
Other: labor dance — The pregnant women and their spouses/partners who wanted to perform the practice were asked to inform the researcher when the labor started. The researcher stayed with the pregnant women and their spouses during the practice and labor process. The pregnant women started to dance with their spouses during the active phase of the labor process accompanied by meditation music in a dim, silent environment. The spouse or partner massaged the pregnant woman's sacral area while dancing.
  Arms: labor dance group

SUMMARY:
ne of the non-pharmacological methods that provide opportunities such as massage and freedom of movement with the support of the spouse / partner is the birth dance.

In order to reduce the pain perceived by the woman and provide emotional support, the birth dance is started in the active phase of the first phase of the labor and continues until the end of the first phase. The woman is given the opportunity to act rhythmically with a relaxing light music with someone she prefers (spouse / partner, mother, midwife, etc.). The hands of the pregnant woman dance in the form of swinging from left to right, on the shoulder of his wife, with music; The partner is massaged by the sacrum area. It is aimed to increase the effectiveness of the method applied by adding spouse / partner support, upright posture and massage in addition to the music and body movements that dance includes, and also to provide emotional support to the woman. In this study, it was aimed to evaluate the effect of birth dance on traumatic birth perception and comfort.

DETAILED DESCRIPTION:
The study was planned as randomized controlled. Pregnant women and their accompanying persons assigned to the study group will be informed about working in the tram room where the pregnant woman is before the active phase begins 'Using the Labor Dance Practice Guide (Annex 3) and cervical dilatation 4 cm. they will be asked to practice in accordance with this guide. Details of the application (such as dance time, rest time) will be recorded in the 'Labor Dance Control Guide' (Annex 4) by the researcher. Pregnant women will be followed by the doctor and midwife responsible for the pregnancy during the tram, and the researcher will not be involved in tram follow-up of the pregnant woman (cervical dilation, pediatric heart sound, contraction follow-up, vital signs of the pregnant woman).

ELIGIBILITY:
Inclusion Criteria:

* Those who were admitted to Hospital for labor
* Those whose cervical dilatation between 4 and 8 cm.

Exclusion Criteria:

* When delivered by cesarean sectio,
* Labor was inducted
* Narcotic analgesics used

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Childbirth Comfort Questionnaire | ten minute after labor dance
  The scale is a five-point Likert type scale with 14 items. In the original of the scale, it is stated that each item can be scored between 1-5 (1 = Strongly disagree, 2 = Mostly disagree, 3 = Partially agree, 4 = Mostly agree, 5 = I totally agree). The minimum score that can be obtained from the scale is 14 and the highest score is 70. The higher the score, the higher the comfort, the lower the lower comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No